CLINICAL TRIAL: NCT07407127
Title: Investigation of Cervical Muscle Endurance and Pressure Pain Threshold in University Students With Temporomandibular Joint Dysfunction: A Case-Control Study
Brief Title: Cervical Muscle Endurance and Pressure Pain Threshold in University Students With TMD: A Case-Control Study
Acronym: TMED-CME-PPT
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, BİNNAZ BOZKURT AKPULAT, Lecturer, Kırıkkale University
Other Study IDs: IGDU-EC-27-03-2024
Record Dates: First submitted 2026-02-01; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Temporomandibular Disorder (TMD); Pain Threshold
Keywords: Temporomandibular joint dysfunction; cervical muscle endurance; pain threshold; posture
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TMD Group: TMD group was defined as scoring 15 points or more on the Fonseca Anamnesis Index (FAI).
- Control Group: Control group was an FAI score below 15.

SUMMARY:
Aim: This study aims to compare the static endurance of cervical region muscles, pressure pain thresholds of selected muscles of the stomatognathic system, and postural characteristics in young adults with and without temporomandibular joint dysfunction (TMD).

Method: A total of 60 university students aged between 18 and 25 years will be included in the study. Participants will be divided into two groups: individuals with temporomandibular joint dysfunction (TMD group, n=30) and healthy controls (control group, n=30). The static endurance of cervical flexor and extensor muscles will be assessed using standardized endurance tests. Pressure pain thresholds of the temporalis, masseter, sternocleidomastoid, and upper trapezius muscles will be measured using a pressure algometer. Postural characteristics will be evaluated using the New York Posture Analysis (NYPA).

DETAILED DESCRIPTION:
The socio-demographic data of the individuals, including age, height, weight, etc., were recorded. The Fonseca Anamnestic Index (FAI) was used to identify the presence of TMD, and individuals with a score above 15 (FAI≥15) were determined to have TMD. Additionally, individuals' muscular endurance was assessed using a standard endurance test, pressure pain thresholds were measured with an algometer, and posture was evaluated using the New York Posture Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled as a student at Igdır University.
* The inclusion criterion for the TMD group was defined as scoring 15 points or more on the Fonseca Anamnesis Index (FAI), while the criterion for the control group was an FAI score below 15.

Exclusion Criteria:

* Underwent surgery in the neck or mandibular regions
* Had a history of intervertebral disk problems, regardless of clinical symptoms
* Experienced mechanical neck pain for ≥3 months
* Had scoliosis
* Had reducible or irreducible displacement of the temporomandibular joint disk
* Had a history of trigeminal neuralgia
* Were undergoing orthodontic dental treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of university students aged 18-25 studying at Igdir University Karaagac Campus.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Cervical Muscle Endurance Assessment | 2 week
  Static endurance of cervical flexor and extensor muscles was measured in seconds. Extensors: participants lay prone, lifted the head slightly, and held a 2-kg weight as long as possible. Flexors: participants lay supine, performed slight craniocervical flexion, and maintained the position. Test ended with pain, loss of position, or sufficient endurance. Intra-observer reliability: flexors 0.71-0.93, extensors 0.73-0.85.
Pressure Pain Threshold Assesment | 2 week
  Pressure pain threshold (PPT) was measured using a Baseline Push-Pull Force Gauge® algometer with a 1 cm rubber tip. After familiarization, pressure was applied perpendicularly to the most sensitive points of the upper trapezius, masseter, temporalis, and SCM muscles until participants reported pain. Each site was tested three times with ≥20 s intervals, and the average value was recorded as the PPT.

SECONDARY OUTCOMES:
Posture Assessment | 2 week
  Posture was assessed using the NYPA, evaluating alignment of 13 body regions including head, neck, shoulders, back, waist, hips, and ankles. Each region was scored 1 (severe impairment), 3 (moderate), or 5 (good), giving a total score of 13-65. Scores were categorized as very good (≥45), good (40-44), moderate (30-39), poor (20-29), or bad (≤19). Reliability coefficients range from 0.93 to 0.98.

CONTACTS AND LOCATIONS:
Overall Officials: Aydan AYTAR, Prof. Dr., Study Director — University of Health Sciences, Gülhane Faculty of Physiotherapy and Rehabilitation; Binnaz Bozkurt Akpulat, MSc., Principal Investigator — Igdir University
Locations (1):
- Igdir University, Iğdır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant confidentiality and because the data were collected solely for the purposes approved by the ethics committee.